CLINICAL TRIAL: NCT06922942
Title: MS-FLOWER: MSCopilot Users' Feedback in Real Life - Outcomes Regarding Integration in Patients' pathWay and Users' ExpeRience
Brief Title: MSCopilot Users' Feedback in Real Life - Outcomes Regarding Integration in Patients' pathWay and Users' ExpeRience
Acronym: MS-FLOWER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADS-MS-FLOWER-2025
Record Dates: First submitted 2025-04-01; First posted 2025-04-11 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Performance of digital tests at home at day 0 (D0), D30, D60, D90, D120, D150 and D180 (Experimental)
  Interventions: Device: MSCopilot Flower mobile application

INTERVENTIONS:
Device: MSCopilot Flower mobile application — MSCopilot Flower includes active tests for walking, cognition, dexterity and vision, and e-questionnaires related to fatigue and Anxiety

SUMMARY:
This US multicenter, prospective cohort study aims to evaluate how MSCopilot can be seamlessly integrated into the current care pathway and identify potential optimizations to enhance its impact on both MS patients and clinicians, facilitating broader implementation. Specifically, the study will assess:

* The overall integration of MSCopilot into routine clinical practice,
* Patients' ability to use MSCopilot at home without supervision,
* The need for patient support when using MSCopilot at home,
* User behavior based on usage analytics data from the MSCopilot mobile app and dashboard,
* Patient adherence to MSCopilot use in routine clinical practice,
* The adequacy of the onboarding/training process for HCPs,
* The effectiveness of HCPs onboarding/training in ensuring successful patient onboarding,
* The variances in user behavior and adherence to MSCopilot use according to socio-demographic factors and EDSS scores

ELIGIBILITY:
Inclusion Criteria:

For patients

* 18 years and older
* With a confirmed and documented MS diagnosis, per the 2010 Revised
* McDonald criteria
* With an EDSS score ranging from 0 to 6.5
* Able to monitor their disease from home (i.e. not hospitalized or under medical assistance).
* Having a personal smartphone with a mobile operating system above 16 for IOS (iPhone) and 8 for Android and having access to a good internet connection.
* Able to read language in which the mobile application is available and able to understand pictograms Having read the information sheet and signed the informed consent form

For HCPs:

* Licensed neurologists trained in the management of Multiple Sclerosis patients and allowed to conduct clinical studies within their departments
* If applicable: nurses or medical assistants specifically trained in the management of Multiple Sclerosis and allowed to participate in clinical studies within their departments
* Ability to use a computer

Exclusion Criteria (for patients):

* Pregnant and nursing women
* Person under guardianship or curatorship
* Inability to use a smartphone application
* Patient who previously participated in a study using MSCopilot

Early termination criteria (for patients):

* exclusion criteria,
* death,
* abandon,
* loss of follow-up,
* investigator's decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
To assess the ease of integrating the MSCopilot dashboard into clinical workflows for neurologists and the ease of use at home for patients with multiple sclerosis. | For neurologists: Day 180 (+/- 30 days) and for patients: Day 1, Day 90 and Day 180 (+/- 30 days)
  Descriptive analysis and acceptance criteria of a minimum score of >2/4 on neurologists' questionnaires regarding the ease of integrating the MSCopilot dashboard into clinical workflows Descriptive analysis and acceptance criteria of a minimum score of >2/4 on patients' questionnaires regarding the ease of use of MSCopilot at home

SECONDARY OUTCOMES:
To assess the integration of MSCopilot dashboard and application into routine clinical practice as well as perceived value for both HCPs and patients. | At Day 180 ± 30days
  Descriptive analysis of neurologists' questionnaires, to be completed after each investigator's last visit, regarding the Health Care Profesionnals (HCPs) dashboard Descriptive analysis and acceptance criteria of a minimum score of >2/4 for each item, of neurologists' questionnaires after the last visit on the HCPs dashboard Descriptive analysis of patients' questionnaires after the last visit regarding MSCopilot app and dashboard use by the HCPs.
  Descriptive analysis and acceptance criteria of a minimum score of >2/4 for each item in patients' questionnaires, to be completed after the follow-up visit, regarding MSCopilot application and dashboard use by HCPs
To assess patients' ability to use MSCopilot at home without supervision. | Day 1 (+/- 30 days)
  Descriptive analysis of patient questionnaires Acceptance criteria of a minimum of >2/4 for each item, of patient questionnaires
To assess patients' ability to use MSCopilot at home without supervision. | Day 90 (+/-30 days)
  Descriptive analysis of patient questionnaires at mid-study Descriptive analysis and acceptance criteria of a minimum score of >2/4 for each item, of patient questionnaires at mid-study
To assess the need for patient support when using MSCopilot at home | Day 180 (+/-30 days)
  Descriptive analysis of nurses or medical assistants' questionnaires (if applicable) Descriptive analysis and acceptance criteria of a minimum score of >2/4 for each item, of nurses or medical assistants' questionnaires (if applicable)
To assess patient adherence to MSCopilot use in routine clinical practice. | Day 1 to Day 180 (+/-30 days)
  Descriptive analysis of the mobile application's adherence data, including:
  Number of performed tests, Number of performed sessions, Number of completed questionnaires.
To assess user behavior based on usage analytics data from the MSCopilot mobile app and the dashboard. | Day 1 to Day 180 (+/-30 days)
  Quantitative analysis of real-world utilization patterns of the MSCopilot mobile app through analytics data Quantitative analysis of real-world utilization patterns of the HCPs dashboard through analytics data
To assess the effectiveness of HCPs onboarding/training in ensuring successful patient onboarding. | At the end of inclusion period (90 days)
  Descriptive analysis of HCPs (neurologists) questionnaires Descriptive analysis and acceptance criteria of a minimum score of >2/4 for each item, of HCPs (neurologists) questionnaires
To assess the effectiveness of HCPs onboarding/training in ensuring successful patient onboarding. | After patient inclusion visit (90 days)
  Descriptive analysis of patient questionnaires Descriptive analysis and acceptance criteria of a minimum score of >2/4 for each item, of patient questionnaires
To assess the adequacy of the onboarding/training process for HCPs, including neurologists, nurses, and medical assistants, focusing on clarity, satisfaction, and confidence in using MSCopilot | After onboarding/training session (Day 0)
  Descriptive analysis of HCPs questionnaires post-onboarding/training session Descriptive analysis and acceptance criteria of a minimum score of >2/4 for each item in HCPs questionnaires post-onboarding/training
To assess the variances in user behavior and adherence to MSCopilot use according to socio-demographic factors and EDSS scores. | Day 1 to Day 180 (+/-30 days)
  Descriptive analysis of how socio-demographic factors and EDSS scores affect patient behavior and adherence to MSCopilot mobile application.
To assess the variances in user behavior and adherence to MSCopilot use according to socio-demographic factors and EDSS scores. | Day 1 to Day 180 (+/-30 days)
  Descriptive analysis of how HCPs socio-demographic factors affect their behavior toward MSCopilot dashboard.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Jenny Feng, New Orleans, Louisiana
  - Robert Naismith, St Louis, Missouri
  - Gabriel Pardo, Oklahoma City, Oklahoma
  - Leorah Freeman, Austin, Texas